CLINICAL TRIAL: NCT02871167
Title: Risk of Infertility Related to Adjuvant Chemotherapy for Early Breast Cancer: Oocyte/Embryo Cryopreservation (CHACRY-1501)
Brief Title: Risk of Infertility Related to Adjuvant Chemotherapy for Early Breast Cancer: Oocyte/Embryo Cryopreservation
Acronym: CHACRY-1501
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: University Hospital, Lille (Other); National Cancer Institute, France (Other Government); University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHACRY-1501; 2016-000808-28 (EudraCT Number); PHRC-K14-010 (Other Grant/Funding Number: INCA)
Record Dates: First submitted 2016-07-28; First posted 2016-08-18 (Estimated); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: oocyte/embryo cryopreservation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oocyte/embryo cryopreservation (Experimental): 1. Controlled ovarian hyperstimulation (COH)
  2. Oocyte/embryo freezing
  Interventions: Procedure: Controlled ovarian hyperstimulation (COH); Procedure: Oocyte/embryo freezing

INTERVENTIONS:
Procedure: Controlled ovarian hyperstimulation (COH) — After information and consent, patients are addressed to a reproductive medicine center.
  The COH will be performed according to a standardized protocol between surgery and the start of adjuvant chemotherapy. Follicular growth will be achieved with an antagonist protocol and by using high dose recombinant FSH (r-FSH). The triggering of the final follicular and oocyte maturation will be obtained by a GnRH (Gonadotropin Releasing Hormone) agonist injection in order to minimize the risk of ovarian hyper-stimulation.
Procedure: Oocyte/embryo freezing — Egg or embryo freezing will be performed according to a standardized protocol: slow-freezing process for embryo; vitrification technique for oocytes. Cryopreserved oocytes and embryos will be stored in the biological bank of each reproductive medicine center (min. 10 years).

SUMMARY:
The aim of the study is to perform a French multicenter prospective interventional study in order to assess the feasibility and safety of ovarian hyperstimulation for oocyte / embryo cryopreservation in young women with breast cancer. The oncologic and reproductive benefit / risk ratio will be investigated in the oncology and reproductive area.

DETAILED DESCRIPTION:
Medical Oncology:

* Information and collection of consent,
* Imaging staging,
* Inclusion
* Physical examination
* Contraception advise given

Reproductive medicine center:

* Ovarian reserve assessment: serum anti-mullerian hormone (AMH) measurement and antral follicle count (AFC) by ultrasound.
* Serology syphilis, hepatitis B and C, HIV (human immunodeficiency virus). In case of embryo cryopreservation, same serology determination for the men.
* Infertility risk and fertility preservation techniques information.
* In case of agreement, this technique will be done during the time-interval between surgery and chemotherapy
* Fertility preservation (COH stimulation, triggering and oocyte retrieval)

Adjuvant chemotherapy:

* The chemotherapy regimen is 3 FEC (fluorouracil epirubicin cyclophosphamide) 100 followed by standard chemotherapy (according to local practice) +/- Trastuzumab. Adjuvant chemotherapy may only begin after the oocyte retrieval.
* Usual adjuvant chemotherapy is not changed

During chemotherapy:

* Clinical exam before each cycle of chemotherapy
* AMH, AFC at cycle 6

After chemotherapy:

* Usual patient monitoring in expert center :

physical examination at Month 3 (M3), M6 M9 M12 M18 and M24 and mammography at M9 then annual

* AMH at Month 3 (M3), M6 M9 M12 M18 and M24
* AFC at Month 12 (M12) and M24

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically proven breast cancer
* Aged 18 to 38 years old
* Planned adjuvant chemotherapy
* No prior chemotherapy
* Affiliated to a public health insurance program
* Informed consent signed by the patient

Exclusion Criteria:

* Metastatic breast cancer
* Planned neo-adjuvant chemotherapy
* Hysterectomy
* Exclusive adjuvant hormonotherapy
* Positive serology for syphilis, hepatitis B or C, or VIH
* Contraindication related to use of r-FSH
* Pregnant or breastfeeding patients

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2034-11 (Estimated)

PRIMARY OUTCOMES:
Quality of oocytes: total number of oocytes preserved | after oocyte retrieval (35-36 hours after triptorelin injection)
  The distribution of the total number of oocytes preserved will be summarized by the mean (standard error) and median (range) and presented with a 95% confidence interval.

SECONDARY OUTCOMES:
Quality of embryos: total number of embryos preserved | at 44-46 hours post intra-cell sperm injection
Type of oocytes | after oocyte retrieval (35-36 hours after triptorelin injection)
  mature, immature, fractured
Toxicity related to the controlled ovarian stimulation according to NCI CTCAE v4.0 scale | 24 months
  Toxicities will be tabulated with frequencies and percentages by type of adverse events and by grade
Serum AMH measurement | baseline, at the end of the first sequence of chemotherapy, at the last injection of treatment, at Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
Antral Follicular Count (AFC) measurement | baseline, at month 3, at month 12, at month 24
Number of Spontaneous or medically assisted pregnancy(ies) | up to 10 years after the end of the study or at 43 years old
  To measure the degree of project completion of subsequent pregnancy(ies)
Rate of patients wishing for re-utilization of their frozen gametes | up to 10 years after the end of the study or at 43 years old
  To assess the number of patients wishing for re-utilization of their frozen gametes
Disease-free survival | through study completion, an average of 5 years
  defined as the interval between inclusion and the first occurrence of local, regional or distant relapse, estimated using the Kaplan-Meier method

OTHER OUTCOMES:
Translational research : circulating nucleic acids quantification: cell-free DNA and microRNAs on blood sample | an average of 6 months
  before 1st cycle of adjuvant chemotherapy, during the adjuvant chemotherapy (end of first sequence), at the end of adjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Maillez, MD, Study Director — Centre Oscar Lambret; Christine Decanter, MD, Study Director — CHRU of Lille - Hôpital Jeanne de Flandre
Locations (28):
- France (28):
  - Hôpital Jean Verdier, Bondy
  - Centre Aliénor d'Aquitaine, Hôpital Pellegrin, Bordeaux
  - CHU de Caen, Caen
  - Centre François Baclesse, Caen
  - Hôpital Antoine Béclère, Clamart
  - Centre Georges François LECLERC, Dijon
  - CHU de Dijon, Dijon
  - CHU REUNION site SUD, La Réunion
  - Centre Oscar Lambret, Lille
  - CHRU Hôpital Jeanne de Flandres, Lille
  - CHU Limoges, Limoges
  - CHU Lyon, Lyon
  - Centre Léon Bérard, Lyon
  - CHU La Conception, Marseille
  - Institut Paoli Calmette, Marseille
  - CHRU Montpellier, Montpellier
  - ICM - Val d'Aurelle, Montpellier
  - CHRU de Nancy, Nancy
  - Institut Curie, Paris
  - Hôpital Cochin, Paris
  - Hôpital TENON, Paris
  - CHU Rouen, Rouen
  - Centre Henri Becquerel, Rouen
  - Institut Curie, Saint-Cloud
  - Hôpital Universitaire de Strasbourg, Strasbourg
  - Oncopole-CHU Toulouse, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No